CLINICAL TRIAL: NCT03590704
Title: Evaluation of Tolerance and Cutaneous Reaction to the Use of Compressive Taping in the Seroma After Surgical Treatment of Breast Cancer
Brief Title: Safety of the Use of Compressive Taping in Seroma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCASafetySeroma
Record Dates: First submitted 2017-10-30; First posted 2018-07-18 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Seroma
Keywords: Taping; Seroma; Safety; Breast Cancer; Physiotherapy
MeSH Terms: conditions — Seroma; Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention Vitaltape® bandage (Experimental): The neuromuscular bandage will be applied after skin antisepsis with 70% alcohol. A 5 cm width Vitaltape® bandage will be used. For the bandage application, a distal base (anchor) with two centimeters of diameter will be maintained with maximum stretching on the seroma and finalized with another base no stretching, of 2 cm, in the proximal region. How many bundles of bandages are required according to the patient's body characteristics and aspect of the flotation region. The bandage will not be applied on the scar. If there are any complications such as itching, redness, discomfort and / or others, the patients will remove the material at home and communicate on return to the institution. They will remain four days approximately for revaluation and intervention suspension.
  Interventions: Device: Vitaltape® bandage

INTERVENTIONS:
Device: Vitaltape® bandage — The neuromuscular bandage will be applied after skin antisepsis with 70% alcohol. A 5 cm width Vitaltape® neuromuscular bandage will be used. For the bandage application, a distal base (anchor) with two centimeters of diameter will be maintained with maximum stretching on the seroma and finalized with another base no stretching, of 2 cm, in the proximal region. How many bundles of bandages are required according to the patient's body characteristics and aspect of the flotation region.

SUMMARY:
Seroma is the most common complication at the beginning of healing after surgery for breast cancer treatment. Its incidence varies in the literature from 2.5 to 90% and is defined as a collection of serous fluid that develops through skin flaps in the dead space after mastectomy or axillary dissection. The physiopathology for seroma formation has not yet been fully understood, but appears to be multifactorial with surgery being the main factor. Although seroma formation is not a threat to life, it can lead to important morbidity due to associated with necrosis, dehiscence, predisposition to sepsis, reduction of shoulder functions due to muscle weakness due to restriction of movement, prolonging the recovery period and, consequently, leading to delay in adjuvant therapy. The best seroma treatment is still not well defined in the literature and the compressive therapy aims to rebalance fluid exchange between the lymphatic system and blood, having as effects the increase of the interstitial pressure, the improvement of the effectiveness of muscular work, increased resistance of the skin and prevention new collection of interstitial fluid. Recently, the Kinesio® Taping method were inserted into clinical practice for its ability to reduce pain and local swelling. Objective: To evaluate the safety of taping in the seroma after surgical treatment of breast cancer. Methodology: This is a pre and post-clinical application of taping on the seroma in women submitted to surgical treatment for breast cancer in the Cancer Hospital III / INCA. The intervention was performed by applying the compression bandage over the seroma region for an average of five days, when the reassessment was performed.

DETAILED DESCRIPTION:
Patients identified by the nursing team with seroma and with indication of aspiration puncture, will be evaluated for eligibility criteria. Those who agree to participate in the study will be assessed and submitted to the intervention on the same day, they will remain with four days approximately for nursing and physiotherapy revaluation for intervention suspension. The neuromuscular bandage will be applied after skin antisepsis with 70% alcohol. A 5 cm width Vitaltape® neuromuscular bandage will be used. For the bandage application, a distal base (anchor) with two centimeters of diameter will be maintained with maximum stretching on the fluctuation region (seroma) and finalized with another base without stretching, of 2 centimeters, in the proximal region. How many bundles of bandages are required according to the patient's body characteristics and aspect of the flotation region. The bandage will not be applied on the scar. If there are any complications such as itching, redness, discomfort and / or others, the patients will remove the material at home and communicate on return to the institution. The interview will be conducted at the entrance to the study, prior to the intervention and the end of the study. In the initial interview will be collected sociodemographic data and life habits. They will be evaluated by questionnaire as the local symptoms caused by the use of the bandages, the tolerance and feeling / referred sensation during and at the end of intervention period, the percentage of seroma volume alteration before and after the use of the bandage, the number of days of use and bandage detachment. All reviews will be carried out by another professional who will not make the interventions. From the hospital record, information will be collected regarding the oncology treatment, histopathological report and clinical data on curative care.

ELIGIBILITY:
Inclusion Criteria:

* Women who developed seroma after surgical treatment for breast cancer, detected by nursing team.

Exclusion Criteria:

* bilateral breast cancer
* neoadjuvant radiotherapy
* wound infection
* reporting of autoimmune diseases (dermatomyositis, hidradenitis suppurativa, nephropathy, lupus erythematosus, morphea, psoriasis, pemphigus vulgaris, scleroderma)
* patients with difficulties of understanding.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Assess dermal changes of using the compressive bandage as a treatment for seroma | 4 to 5 days
  Dermal changes were evaluated at the site of application of the bandage of the 35 participants, such as discoloration, local temperature increase, skin peeling, presence of wound and formation of bullous lesions at the site of application of neuromuscular bandage, graded in mild, moderate or severe , according to the severity of the change, from a semi-structured questionnaire.

SECONDARY OUTCOMES:
Seroma volume difference | 4 to 5 days
  It was verified from the comparison between the volumes of liquid punctured by nursing punctured by the nursing team on the day of application and on the return of the patient
It was evaluated the patient's tolerance to the use of compressive bandages | 4 to 5 days
  It was counted how many of the 35 patients felt pain, itching, burning, discomfort, tightness, increased fluctuation (seroma) at the place where the bandage was applied. The symptoms were graded according to the Visual Numeric Scale (0-10), where 0 was considered to be sensations and 10 was unbearable sensation with the use of bandages.
It was evaluated the patient satisfaction with the use of compressive bandages | 4 to 5 days
  It was evaluated how many of the 35 participants were satisfied with the use of the bandage, being graded according to the Visual Numerical Scale, where 0 was considered totally dissatisfied and 10 was totally satisfied.
It was assessed whether the patient felt secure with compressive bandage | 4 to 5 days
  It was evaluated how many of the 35 participants felt safe using the bandage. For each participant, safety was graded according to the Visual Numerical Scale, where 0 was considered totally dissatisfied and 10 was completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Fabro, Master, Principal Investigator — INCA - Brazil
Locations (1):
- Erica Alves Nogueira Fabro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Fabro EAN, Teodozio CGC, Costa RM, Macedo FO, Cardoso ACDDLM, Jacob RBE, Thuler LCS, Bergmann A. Clinical Experience with Compression Taping to Treat Seroma After Breast Cancer Surgery: A Medical Device Clinical Study. Adv Skin Wound Care. 2022 Jul 1;35(7):1-6. doi: 10.1097/01.ASW.0000831068.34587.3d. PMID 35723961